CLINICAL TRIAL: NCT05717998
Title: A Pilot Study to Evaluate Early Signs of Myocardial Injury After Thoracic Radiotherapy Using Imaging and Blood-Based Biomarkers
Brief Title: Imaging and Blood-Based Biomarkers for the Evaluation of Early Signs of Myocardial Injury After Thoracic Radiation Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Eric Miller, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-20351; NCI-2021-08714 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-09-02; First posted 2023-02-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Lung Non-Small Cell Carcinoma; GastroEsophageal Cancer; Esophagus Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-correlative (CMR, PET/CT, biospecimen collection): Within 2 weeks of starting RT, patients undergo CMR, cardiac PET/CT and blood sample collection at baseline, then between fractions 12-17 of RT and at 6 months after completion of RT.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging of the Heart; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection
Procedure: Computed Tomography — Undergo cardiac PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging of the Heart — Undergo CMR
  Other Names: Cardiac MRI; Heart MRI
Procedure: Positron Emission Tomography — Undergo cardiac PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This study assesses for early signs of damage to the heart following chest radiation therapy using both imaging (cardiac magnetic resonance imaging and cardiac positron emission tomography) and changes in blood biomarkers. This study determines if any changes in the heart muscle can be detected either during the course of radiation therapy or shortly thereafter using specialized imaging techniques or blood tests. Cardiac magnetic resonance imaging may be used to help provide information about changes in the heart structure and function following radiation therapy. Positron emission tomography looks at differences in how the heart takes up radioactive sugar which is injected into the vein to assess changes in heart function following radiation therapy. This study may help identify patients at risk of heart issues following radiation therapy to the chest and ultimately help in the development of more effective and safe treatments for cancer in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate and quantitate early changes in myocardial fibrosis following thoracic radiation therapy (RT).

II. To assess quantitative early changes in myocardial inflammation after thoracic RT.

III. To determine if thoracic RT is associated with early changes in myocardial metabolism as assessed with cardiac positron emission tomography (PET).

SECONDARY OBJECTIVES:

I. To evaluate and quantitate early changes in subclinical myocardial dysfunction after thoracic RT.

II. To determine if thoracic RT is associated with early changes in myocardial metabolism using alternative cardiac PET-derived biomarkers.

III. To evaluate and quantitate early changes in blood-based biomarkers after thoracic RT.

IV. To assess the incidence and severity of cardiac events following completion of thoracic RT.

OUTLINE:

Within 2 weeks of starting RT, patients undergo cardiac magnetic resonance (CMR) imaging, cardiac positron emission tomography (PET)/computed tomography (CT) and blood sample collection at baseline, then between fractions 12-17 of RT and at 6 months after completion of RT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been evaluated by a radiation oncologist and have been felt to be suitable to undergo thoracic RT for histologically confirmed NSCLC with a dose range of 60-70 Gy at 1.8-2 Gy per fraction OR histologically confirmed clinical stage I-IVA (AJCC 8th ed) middle or thoracic esophageal or gastroesophageal cancer (squamous cell carcinoma or adenocarcinoma) with a planned dose range of 41.4-60 Gy at 1.8-2 Gy per fraction as part of treatment of their malignancy
* Concurrent chemotherapy is permitted
* For NSCLC patients, both concurrent and/or adjuvant immunotherapy is permitted
* Patients participating in other research studies are eligible as long as participation in this study does not interfere with activities required in the other studies
* Patients with no contra-indications to magnetic resonance (MR) or PET imaging as stated in the section exclusion criteria
* For the delayed enhancement and the T1 contrast mapping portions of the study, the patient must have an adequate baseline renal function defined as an estimated glomerular filtration rate (eGFR) > 30 ml/min per the Ohio State Institutional Guidelines. Of note, if the patient's eGFR is =< 30 ml/min, the patient would still be eligible for enrollment, but only the strain-encoded (SENC) imaging and T2 mapping non-contrast sequences would be obtained. The dynamic contrast-enhanced (DCE) and T1 mapping sequences, which require intravenous (IV) contrast, would not be included
* Patients with moderate to end-stage renal disease, or who are at high-risk of nephrogenic systemic fibrosis (e.g. hepatorenal syndrome, liver transplant, acute renal failure, chronic kidney disease, and iron overload conditions) would still be eligible for enrollment, but only the non-contrast SENC and T2 mapping imaging sequences would be obtained. The DCE and T1 mapping sequences, which require IV contrast, would not be included
* Age >= 18 years old
* Within 4 weeks of study entry: patients must have vital signs, history/physical examination, and kidney function test (eGFR)
* Ability to provide written informed consent obtained prior to participation in the study and any study specific procedures being performed
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test within 14 days of the study entry. Urine human chorionic gonadotropin (HCG) is an acceptable pregnancy assessment

Exclusion Criteria:

* Subjects who are breast-feeding, or have a positive pregnancy test will be excluded from the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Medical contraindications to MR imaging (e.g. pacemakers, metallic implants, aneurysm clips, known contrast allergy to Gadolinium contrast, pregnancy, nursing mothers, weight greater than 350 pounds)
* Subjects with advanced renal disease (eGFR < 45 mL/min/1.72m^2) - exclusion from receipt of contrast, but may still be enrolled for basic CMR imaging (left ventricular ejection [LVEF], strain, T2, etc)
* Medical contraindications to PET imaging (e.g. pregnancy, nursing mothers, weight greater than 420 pounds - scanner limit)
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other condition that could prevent compliance with study procedures or providing informed consent
* Subjects who are prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suitable to undergo thoracic RT for histologically confirmed non-small cell lung cancer (NSCLC) OR histologically confirmed clinical stage I-IVA (American Joint Committee on Cancer [AJCC] 8th edition [ed]) middle or thoracic esophageal or gastroesophageal cancer (squamous cell carcinoma or adenocarcinoma) at Ohio State University Comprehensive Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Changes in extracellular volume (ECV) | Baseline up to 6 months post-radiation therapy (RT)
  To identify the presence of cardiac fibrosis as assessed by cardiac magnetic resonance-derived ECV during and shortly after RT.
Changes in myocardial T2 | Baseline up to 6 months post-RT
  To identify the presence of cardiac magnetic resonance-derived cardiac inflammation using T2 mapping during and shortly after RT.
Changes in myocardial metabolism | Baseline up to 6 months post-RT
  To identify changes in myocardial metabolism measured as standardized uptake value (SUV) max during and shortly after RT using myocardial PET.

SECONDARY OUTCOMES:
Blood-based biomarkers | Baseline up 6 to months post-RT
  Biomarkers including serum troponin, N-terminal Pro Brain-type Natriuretic Peptide (NT-proBNP), C-reactive protein, carboxy-terminal propeptide of procollagen type I (PICP), and amino-terminal propeptide of procollagen type I (PINP) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Miller, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu